CLINICAL TRIAL: NCT05824377
Title: To Determine the Best Feeding Practice in Preterm Infants on Non-invasive Ventilation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rajeev Kumar (Other Government)
Responsible Party: Sponsor-Investigator, Rajeev Kumar, Principal Investigator, Cook County Health
Organization: Cook County Health (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 22-058
Record Dates: First submitted 2023-03-28; First posted 2023-04-21 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Prematurity; Extreme; Feeding Patterns; Ventilator Lung; Newborn
Keywords: Preterm infants; Feeding methods; bolus feeds; continuous feeds; non-invasive ventilation; RAM cannula
MeSH Terms: conditions — Premature Birth; Feeding Behavior; Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: Infants will be randomized into 2 groups; one will receive continuous nasogastric feeding and the other group will receive intermittent bolus feeds.
  Each group will be stratified as per weight, thus (<1000 g, 1000-1500 g, and > 1500 g). It will be 1-1 randomization and will be randomized into each group by pulling a sealed envelope. Protected Health Information (PHI) will be de-identified by assigning a study code.
  Sample size: A sample size of at least 23 in each arm was calculated using the SAS system. A power of 80% and a mean difference of 40% decrease in the length of time to achieve full feeds; and an SD of 8.5 was considered while calculating the number of patients. The mean length of time to achieve full feeds in our NICU as per chart review was 17 +/- 8.5 days.
Who Masked: Outcomes Assessor
Masking Description: Caregivers, study personnel and nurses will not be blinded, as blinding will be hard for the treating team. Parents will not be blinded as we inform about the infant's progress and plan routinely. Statisticians will be blinded during (they will receive de-identified data).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus Feeding (Experimental): Intermittent bolus feeding will be defined as delivering enteral nutrition multiple times, usually every 2-3 hours over 15 - 30 minutes by gravity or an electric pump.
  It will be further stratified as per weight ( less than 1000 g, 1000-1500 g, >1500 g).
  Interventions: Other: Intermittent Bolus Feeds
- Continuous Feeding (Experimental): Continuous feeding will be defined as delivering enteral nutrition with constant speed for 24 hours via a nutritional pump.
  It will be further stratified as per weight ( less than 1000 g, 1000-1500 g, >1500 g).
  Interventions: Other: Continuous Feeds

INTERVENTIONS:
Other: Continuous Feeds — Continuous feeds will be delivered via an indwelling nasogastric/orogastric tube with a continuous infusion pump.
  Arms: Continuous Feeding
Other: Intermittent Bolus Feeds — Intermittent bolus feedings will be given by gravity every 3 hours over 15- 30 minutes.
  Arms: Bolus Feeding

SUMMARY:
To evaluate the duration to reach full feeds by comparing continuous gavage feeds versus bolus feeds in preterm infants who are on non-invasive respiratory support (RAM cannula - short binasal prongs).

DETAILED DESCRIPTION:
Methods:

The study will be a randomized control trial at our NICU (Neonatal Intensive Care Unit) (Level III). Preterm infants on non -invasive ventilation (nasal intermittent positive pressure ventilation (NIPPV)/ continuous positive airway pressure (CPAP)) will be randomly assigned into either continuous feeds or bolus feeds groups. Baby will be fed enterally through a nasogastric tube via continuous or bolus feeds using either maternal milk or formula, according to parental choice. Feeds will be advanced as per the feeding guidelines or per treating physician. Currently we use both bolus and continuous feeding practice in our NICU, as per physician's discretion.

Intervention:

Infants will be randomized into 2 groups; one will receive continuous nasogastric feeding and the other group will receive intermittent bolus feeds. Continuous feeds will be delivered via an indwelling nasogastric/orogastric tube with a continuous infusion pump. Intermittent bolus feedings will be given by gravity every 3 hours over 15- 30 minutes.

Parents' consent will be taken when the infant is qualified for the study. The consent will be taken by one of the coinvestigators. Each coinvestigator will be trained to consent for standardization. Non-English-speaking parents will be consented using the medical video interpreter (Voyce). Accent will not be obtained as neonates aren't mature to give accent.

Patients will be randomized into each group by pulling a sealed envelope.

Monitoring for complications:

During the study, infants will be monitored for any complications due to either feeding protocol like feeding intolerance, reflux, abdominal distension, poor weight gain, any risk of aspiration pneumonia or necrotizing enterocolitis (NEC). Such symptoms are usually monitored by our NICU team as per our guidelines. These feeding issues can be encountered in either group. If such problems are encountered, feeding protocol will be changed as per the physician's clinical decision. Parents will be informed of the changes. Intention to treat protocol will be used while calculating the statistical analysis.

Guidelines for withholding the feeds (bolus or intermittent) or changing either group will be:

1. Excessive gastric residual (> 50% of the volume fed)
2. Increase in abdominal girth (>1.5-2.5 cm along with other signs and symptoms of intolerance to feeds)
3. Poor/slow weight gain (rate of weight gain is significantly below that expected for age and sex, or if weight has dropped ≥2 major percentile lines)
4. Occult blood positive in stools/visible blood in the stools
5. Concerns for neonatal sepsis clinically as per attending's discretion
6. Apnea pertaining for more than 20 secs alone or apnea for > 10 seconds along with bradycardia (<80) or desaturations (hypoxemia as per gestational age); and occurring more than 2 or 3 times a day and requiring intervention
7. Abnormal Abdominal X rays concerning for suspected NEC or NEC as per Bell's criteria
8. Infants who need to be on invasive ventilation
9. Treating physician's clinical decision

Feeding protocol:

BW: 500 -1000 grams:

Initiate: When baby is stable. Start with trophic feeds, that is, 5 -10 ml/kg/day.

Advance: If tolerating trophic feeds for 2-3 days, advance feeds by 10 ml/kg/day.

Initial choice of milk: Breast Milk/Donor Breast Milk / Formula (Enfamil) - 20Kcal/Oz.

Fortify: When 60-80 ml/kg/day feeds are reached, fortify to 22Kcal/Oz and within next few days to 24 Kcal/Oz.

BW 1000 - 1500 grams:

Initiate: When baby is stable. Trophic feeds 5-10 ml/kg/day. Advance: 15-20 ml/kg/day Initial choice of milk, fortifying and full feeds as above.

BW 1500 grams and above:

Initiate: 30 ml/kg/day. Advance: 20 -35 ml/kg/day Initial choice of milk, fortifying and full feeds as above.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm Infants 24- 34 weeks of gestation
2. On Non-invasive ventilation (NIPPV/CPAP/HFNC)
3. Nothing by mouth (NPO) or on trophic feeds (<20 ml/kg/day) at the time of randomization.

Exclusion Criteria:

1. Gestational Age > 34 weeks
2. Infants on invasive ventilation or low flow nasal cannula and on feeding volume more than trophic feeds.
3. Major congenital anomalies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Day of life to reach full feeds | From the date of randomization until the date of NICU discharge/death, assessed up to 1 year.
  the day of life to reach full feed, that is, 120 ml/kg/day.

SECONDARY OUTCOMES:
Feeding interruptions | From the date of randomization until the date of NICU discharge/death, assessed up to 1 year.
  Interruptions while feeding, which includes NPO days, Lab usage and Radiological evaluation.
Time to reach (day of life) first oral feed | From the date of randomization until the date of NICU discharge/death, assessed up to 1 year.
  Day of life when infant was taking oral feeds (no feeds by nasogastric tube)
Weight gain, head circumference (HC) and Length. | From the date of randomization until the date of NICU discharge/death, assessed up to 1 year.
  Anthropometric parameters
Length of hospital stay | From the date of randomization until the date of NICU discharge/death, assessed up to 1 year.
  Total duration of hospital stay
Use of investigative medicine for feeding intolerance | From the date of randomization until the date of NICU discharge/death, assessed up to 1 year.
  Use of radiographic imaging or blood work-up to rule out any feeding intolerance

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Kumar, MD, Principal Investigator — Cook County Health
Locations (1):
- Cook County Helath, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cresi F, Maggiora E, Borgione SM, Spada E, Coscia A, Bertino E, Meneghin F, Corvaglia LT, Ventura ML, Lista G; ENTARES Study Research Group. Enteral Nutrition Tolerance And REspiratory Support (ENTARES) Study in preterm infants: study protocol for a randomized controlled trial. Trials. 2019 Jan 18;20(1):67. doi: 10.1186/s13063-018-3119-0. PMID 30658676
- [Background] Wang Y, Zhu W, Luo BR. Continuous feeding versus intermittent bolus feeding for premature infants with low birth weight: a meta-analysis of randomized controlled trials. Eur J Clin Nutr. 2020 May;74(5):775-783. doi: 10.1038/s41430-019-0522-x. Epub 2019 Oct 28. PMID 31659243
- [Background] Mukerji A, Abdul Wahab MG, Razak A, Rempel E, Patel W, Mondal T, Beck J. High CPAP vs. NIPPV in preterm neonates - A physiological cross-over study. J Perinatol. 2021 Jul;41(7):1690-1696. doi: 10.1038/s41372-021-01122-6. Epub 2021 Jun 5. PMID 34091605
- [Background] Premji SS, Chessell L. Continuous nasogastric milk feeding versus intermittent bolus milk feeding for premature infants less than 1500 grams. Cochrane Database Syst Rev. 2011 Nov 9;2011(11):CD001819. doi: 10.1002/14651858.CD001819.pub2. PMID 22071802
- [Background] Dumpa V, Kamity R, Ferrara L, Akerman M, Hanna N. The effects of oral feeding while on nasal continuous positive airway pressure (NCPAP) in preterm infants. J Perinatol. 2020 Jun;40(6):909-915. doi: 10.1038/s41372-020-0632-2. Epub 2020 Feb 21. PMID 32086439
- [Background] Akintorin SM, Kamat M, Pildes RS, Kling P, Andes S, Hill J, Pyati S. A prospective randomized trial of feeding methods in very low birth weight infants. Pediatrics. 1997 Oct;100(4):E4. doi: 10.1542/peds.100.4.e4. PMID 9310537